CLINICAL TRIAL: NCT01225484
Title: Perioperative Analgetic Therapy After Knee Arthroplasty
Brief Title: Perioperative Analgesia After Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Landeskrankenhaus Feldbach (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Karl Trauner, M.D., Landeskrankenhaus Feldbach
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-315 ex 09/10
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Knee Arthroplasty
Keywords: Knee arthroplasty, perioperative analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CFNB, periarticular infiltration (Active Comparator)
  Interventions: Procedure: Continuous femoral nerve block + periarticular infiltration
- Intraarticular catheter, periarticular infiltration (Active Comparator)
  Interventions: Procedure: Continuous femoral nerve block + periarticular infiltration; Procedure: Intraarticular and periarticular ropivacaine

INTERVENTIONS:
Procedure: Continuous femoral nerve block + periarticular infiltration — Initial bolus of ropivacaine 5mg/ml 30mls into the femoral-nerve-catheter preoperatively. Periarticular infiltration of ropivacaine 2mg/ml 150 mls intraoperatively. Continuous perineural infusion of ropivacaine 2mg/ml at a rate of 6 mls/hr postoperatively. Rate can be adjusted to achieve optimal pain control and avoid motor blockade.
  Other Names: CFNB plus periarticular infiltration
Procedure: Intraarticular and periarticular ropivacaine — Periarticular infiltration of 150 mls ropivacaine 2mg/ml intraoperatively, intraarticular injection of 40 mls ropivacaine 2 mg/ml at skin closure followed by infusion of ropivacaine 2 mg/ml at a rate of 4 mls/hr delivered by an intraarticular catheter until the morning of postoperative day 3.
  Other Names: Intraarticular ropivacaine plus periarticular ropivavaine
  Arms: Intraarticular catheter, periarticular infiltration

SUMMARY:
The purpose of this study is to compare two accepted methods of pain control in knee arthroplasty surgery.The first method combines the periarticular injection of ropivacaine with continuous blockade of the femoral nerve.The second method uses periarticular infiltration of ropivacaine in combination with an bolus of ropivacaine into an intraarticular catheter placed intraoperatively followed by a continuous intraarticular infusion of ropivacaine. All patient will also receive a sustained-release oral opioid and oral rescue opioids determined by pain severity using the Visual Analog Scale (VAS)

ELIGIBILITY:
Inclusion Criteria:

* Elective primary knee arthroplasty
* ASA I,II,&III patients
* Spinal Anaesthesia

Exclusion Criteria:

* Patients refusing consent
* Contraindications to regional anaesthesia
* Preexisting neurological disease
* Alcohol or drug abuse
* Inability to use the outcome assessment tools
* Wheel chair or walker dependent
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Static and dynamic pain scores (VAS) | 72 h

SECONDARY OUTCOMES:
Maximum knee flexion (active/passive)>= 90° | 72 h

CONTACTS AND LOCATIONS:
Overall Officials: Karl Trauner, M.D., Principal Investigator — LKH Feldbach
Locations (1):
- LKH Feldbach, Feldbach, Austria